CLINICAL TRIAL: NCT03912129
Title: Autoimmune Cytopenia: Genetics and Pathophysiological Mechanism in Pediatric Evans Syndrome
Acronym: ACTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut des maladies génétiques, Paris (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2018/49
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Evans Syndrome
Keywords: pediatric Evans Syndrome; genetic causes; immunophenotyping immunologic explorations
MeSH Terms: conditions — Evans Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pediatric Evans Syndrome (Other): Collection of biological samples of children with pSE included in the the OBS'CEREVANCE cohort and their parents, for genetic and functional immunological analyzes.
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample — A first systematic approach by Targeted-Next Generation Sequencing will be used on the entire cohort of patients with pSE. This step will be performed on a sequencing chip specifically developed to detect anomalies in known genes involved in autoimmunity.
  In patients for whom no mutations are identified, a whole exome sequencing (WES) approach will be applied to patients and their parents to seek to identify mutations in new genes that may be related to pSE.
  In patients for whom this WES approach is unsuccessful, the search for somatic lymphocyte mutations, or copy number variants will be performed before considering a complete genome sequencing .
  If several candidate genes are identified, the clinical data provided by the CEREVANCE and the phenotypic analyses carried out prior to genetic analyses by the CEDI laboratory will guide the choices to prioritize the study of the identified variants.

SUMMARY:
Characterization of the genetic causes, and of the immunopathological clinical and biological manifestations in children with pediatric Evans syndrome included in a prospective national observational cohort of rare diseases.

DETAILED DESCRIPTION:
Pediatric Evans syndrome (pES) is a rare and severe disease combining immunologic thrombocytopenic purpura (ITP) and autoimmune hemolytic anemia (AIHA). French patients from the 30 hematologic pediatric centers are from 2004 included in a prospective national OBS'CEREVANCE cohort.

A first pilot study revealed a monogenic cause in 7/18 patients (40%) with mutations in the CTLA-4, LRBA, STAT3 GOF, and KRAS. TNGS or exome studies were performed between 2015 and 2018 inn 80 patients with pSE from the OBS'CEREVANCE cohort. This approach, combined with by immunophenotyping lymphocyte, identified a genetic cause of the disease in 26 patients (32%) (TNFRSF6, CTLA4, LRBA, STAT3 GOF, PIK3CD, RAG1, KRAS) and potential causal mutations in 18 other patients (22%), bringing the proportion of potential single gene cause to 76%.

The central hypothesis of this study is that most, if not all, cases of pSE are related to a monogenic or digenic cause, possibly with the intervention of genetic modifiers such as somatic mutations.

ELIGIBILITY:
Inclusion Criteria:

* Patient registered in the French national prospective OBS'CEREVANCE cohort
* Diagnosis of pediatric Evans syndrome (PTI+AHAI)
* Age strictly under 18 years at the initial onset
* Child residing in metropolitan France and affiliated to a french health insurance system
* Free, informed, written and signed consent

Exclusion Criteria:

* Evans syndrome secondary to chemotherapy, bone marrow transplantation or organ transplantation.
* Refusal to participate from parents/patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-05-06 (Estimated); Primary Completion 2022-05-06 (Estimated); Study Completion 2022-05-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients for whom a causal mutation has been identified (known or new) | after the genetic analyzes carried out on all the participants included, may 2022
The number of biological samples collected for PSE children included in the OBS'CEREVANCE cohort and their relatives will be recorded | every 3 months, between may 2019 and may 2022

SECONDARY OUTCOMES:
Immunopathological clinical manifestations | after the genetic analyzes carried out on all the participants included, may 2022
Abnormalities of lymphocyte immunophenotyping | after the genetic analyzes carried out on all the participants included, may 2022
The correlation between causal mutations identified with the clinical and immunological phenotype | after the genetic analyzes carried out on all the participants included, may 2022
Physiopathological and potentially therapeutic classification of pES-T | after the genetic analyzes carried out on all the participants included, may 2022